CLINICAL TRIAL: NCT02176876
Title: A Phase 1b, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GS-5745 in Subjects With Rheumatoid Arthritis
Brief Title: Safety, Tolerability, and Pharmacokinetics of GS-5745 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-373-1276; 2013-005396-41 (EudraCT Number)
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; RA; GS-5745; MMP9; phase 1
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — andecaliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GS-5745 (Experimental): Participants will receive GS-5745 every 2 weeks for a total of 3 infusions.
  Interventions: Drug: GS-5745
- Placebo to match GS-5745 (Placebo Comparator): Participants will receive placebo to match GS-5745 every 2 weeks for a total of 3 infusions.
  Interventions: Drug: Placebo to match GS-5745

INTERVENTIONS:
Drug: GS-5745 — GS-5745 400 mg administered intravenously
  Arms: GS-5745
Drug: Placebo to match GS-5745 — Placebo to match GS-5745 administered intravenously
  Arms: Placebo to match GS-5745

SUMMARY:
This study is to assess the safety, tolerability, and pharmacokinetics (PK) of multiple infusions of GS-5745 in adults with rheumatoid arthritis (RA). Participants will be randomized in a 4:1 ratio to receive 1 intravenous (IV) infusion of GS-5745 or placebo every 2 weeks, for a total of 3 IV infusions.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age, inclusive, at time of screening
* Weight: ≥ 45 to < 120 kg
* Males or non-pregnant, non-lactating females
* Diagnosis of RA according to the 1987 revised American College of Rheumatology (ACR) for the classification of RA
* Active disease, defined as a mean high sensitivity C-reactive protein (hsCRP) value from Visits 1 & 2 of ≥ 8 mg/L
* Individuals taking chronic Disease-Modifying Antirheumatic Drugs (DMARDs) should be on a stable dose for at least 45 days prior to randomization
* Chronic use of systemic corticosteroids up to a maximum of 10 mg/day of prednisone or equivalent is allowed if dose is stable for at least 30 days prior to randomization
* Nonsteroidal Anti-inflammatory Drugs (NSAIDs) or other analgesics are allowed if doses are stable for at least 30 days prior to randomization

Exclusion Criteria:

* Have a document medical history of anaphylaxis
* Positive HIV antibody during screening
* Positive hepatitis B surface antigen (HBsAg), or positive hepatitis B core antigen (HBcAg), followed by a positive hepatitis B virus (HBV) DNA by quantitative polymerase chain reaction (PCR) during screening
* Positive hepatitis C virus (HCV) antibody followed by a positive HCV viral RNA during screening
* A positive QuantiFERON-tuberculosis (TB) GOLD test during screening
* History of malignancy within the last 5 years except for individuals who have been treated locally for non-melanoma skin cancer or cervical carcinoma in situ
* Severe dementia or Alzheimer's disease, chronic medical or psychiatric problem, or alcohol or drug abuse, that in the judgment of the investigator may interfere with individual's ability to comply with study procedures
* Any serious cardiac event such as myocardial infarction, unstable or life-threatening arrhythmia, hospitalization for cardiac failure within 6 months prior to randomization or any significant or new ECG finding at Visit 1 as judged by the investigator
* History of significant systemic involvement secondary to RA such as vasculitis, pulmonary fibrosis, or Felty's syndrome
* History of or current inflammatory joint disease, other than RA, such as gout, reactive arthritis, psoriatic arthritis, seronegative spondylarthritis, or Lyme disease
* History of or current autoimmune or rheumatic disorders, other than RA, such as systemic lupus erythematosus, inflammatory bowel disease, fibromyalgia, polymyalgia rheumatic, scleroderma, inflammatory myopathy, mixed connective tissue disease, or other overlap syndrome
* Any chronic medical condition (including, but not limited to, cardiac or pulmonary disease) that, in the judgment of the investigator, would make the individual unsuitable for the study or would prevent compliance with the study protocol
* Treatment with antibiotics for a clinical infection or other medical condition within 30 days prior to randomization
* Treatment with azathioprine or cyclosporine 90 days prior to randomization
* Treatment with infliximab, golimumab, adalimumab, abatacept, tocilizumab within 90 days; and etanercept or anakinra within 30 days of randomization
* Treatment with rituximab or any B-cell depleting agent within 12 months of randomization
* Treatment with any other marketed or investigational biologic within 5 half-lives of the molecule or if unknown within 90 days of randomization
* Administration of any investigational drug or use of any investigational device within 30 days prior to randomization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, changes in laboratory tests and vital signs from baseline, and development of immunogenicity after dosing | Up to 100 days
  This composite endpoint will measure the safety and tolerability profile of GS-5745.

SECONDARY OUTCOMES:
PK profile of GS-5745 | Pre-infusion, 30 minutes, 4 hours, and 24 hours post-infusion on Day 1; pre-infusion and 30 minutes post-infusion on Days 15 and 29; Days 4, 8, 36, and 43
  This composite endpoint will measure the plasma PK profile of GS-5745. The following parameters will be measured, where applicable:
  * Cmax: maximum observed concentration of drug in plasma
  * Tmax: time of Cmax
  * Clast: last observable concentration of drug
  * Tlast: time of Clast
  * AUClast: concentration of drug from time zero to the last quantifiable concentration
  * AUCinf: concentration of drug extrapolated to infinite time (area under the plasma concentration versus time curve extrapolated to infinite time)
  * AUCtau: concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval)
  * Ctau: observed drug concentration at the end of the dosing interval
  * λz: terminal elimination rate constant
  * CL: systemic clearance of the drug following intravenous administration
  * Vz: volume of distribution of the drug following intravenous administration

CONTACTS AND LOCATIONS:
Overall Officials: David Gossage, MD, Study Director — Gilead Sciences
Locations (4):
- Prague, Czechia
- Hungary (3):
  - Balatonfüred, Veszprém megye
  - Budapest
  - Debrecen

REFERENCES:
- [Derived] Gossage DL, Cieslarova B, Ap S, Zheng H, Xin Y, Lal P, Chen G, Smith V, Sundy JS. Phase 1b Study of the Safety, Pharmacokinetics, and Disease-related Outcomes of the Matrix Metalloproteinase-9 Inhibitor Andecaliximab in Patients With Rheumatoid Arthritis. Clin Ther. 2018 Jan;40(1):156-165.e5. doi: 10.1016/j.clinthera.2017.11.011. Epub 2017 Dec 26. PMID 29287749